CLINICAL TRIAL: NCT00378820
Title: The Effect of Whey and Casein With and Without Milk Minerals on IGFs in Prepubertal Boys
Brief Title: The Effect of Whey and Casein on IGFs in Prepubertal Boys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: ARLA Ingredients a.m.b.a. (Unknown)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: KF 01-072/04; D-111
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2006-09

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Children; Whey; Casein; Milk minerals; Growth factors; IGF-I; Insulin
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Insulin Resistance | interventions — Whey; Caseins

INTERVENTIONS:
Behavioral: Whey without milk minerals
Behavioral: Whey with milk minerals
Behavioral: Casein without milk minerals
Behavioral: Casein with milk minerals

SUMMARY:
It is not clear which milk compounds are responsible for the growth stimulation. Through short term intervention studies in prepubertal children, we will test the effects of whey, casein, and milk minerals (especially Ca/P). Outcomes will be IGF-I, IGFBP-3, p-amino acids, oral glucose tolerance test (insulin, glucose, GLP-1 and 2, C-peptide, proinsulin) and markers for bone turn-over in blood and urine (s-osteocalcin, s-bone alkaline phosphatase, urine Dpyr, Ntx) as well as blood pressure.

DETAILED DESCRIPTION:
Milk has evolved to support high growth velocity in newborns and observational and intervention studies suggest that milk has special growth stimulating properties especially regarding body size, bone mass and gut. We have previously shown that a one week high-dose intervention with milk, but not meat, increased fasting IGF-I and insulin levels in prepubertal boys. It is not clear which milk compounds are responsible for the growth stimulation. Through short term intervention studies in prepubertal children, we will test the effects of whey, casein, and milk minerals (especially Ca/P). Outcomes will be IGF-I, IGFBP-3, p-amino acids, oral glucose tolerance test (insulin, glucose, GLP-1 and 2, C-peptide, proinsulin) and markers for bone turn-over in blood and urine (s-osteocalcin, s-bone alkaline phosphatase, urine Dpyr, Ntx) as well as blood pressure. Exploring the growth stimulating effects of these milk components will improve the understanding of dietary effects on growth and bone metabolism, and will be valuable for the diary industry developing dietary products supporting growth e.g. infant formula, products for clinical nutrition and milk based products for nutritional rehabilitation of malnourished children in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* habital milk intake:200 - 500 mL/d

Exclusion Criteria:

* chronic illnesses
* children who suffer from any condition likely to affect their protein metabolism or growth

Ages: 8 Years to 8 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2004-07; Study Completion 2005-04

PRIMARY OUTCOMES:
IGF-I
IGFBP-3
Insulin
Glucose

SECONDARY OUTCOMES:
Blood Pressure
Body Composition
Adiponectin
Leptin
Ghrelin
C-peptide
OGGT
Urea Nitrogen
Amino Acids
Osteocalcin
BAP
CTX

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, Dr Med Sci, Study Chair — Institute of Human Nutrition, Rolighedsvej 30, DK-1958 Frederiksberg C, Denmark
Locations (1):
- Institute of Human Nutrition, Rolighedsvej 30, Frederiksberg C, Denmark